CLINICAL TRIAL: NCT00662636
Title: Phase I Trial of the Combination of Dasatinib and Lapatinib
Brief Title: Dasatinib and Lapatinib Ditolsylate in Treating Patients With Advanced Solid Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0616; NCI-2009-01197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0616 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Dasatinib; Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive oral dasatinib and lapatinib ditosylate once daily on days 1-28.
  Interventions: Drug: dasatinib; Drug: lapatinib ditosylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: pharmacological study — Correlative study (cohort II only)
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative study (cohort II only)

SUMMARY:
RATIONALE: Dasatinib and lapatinib ditoslylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of dasatinib and lapatinib ditoslylate when given together in treating patients with advanced solid tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose of dasatinib combined with lapatinib.

II. To describe the toxicities associated with this treatment combination. III. To assess the pharmacokinetic interaction of lapatinib and dasatinib. IV. To assess the effect of the lapatinib and dasatinib combination on circulating tumor cells and on osteoclast precursor activation.

V. To study the association of clinical (toxicity and/or tumor response or activity) with the pharmacokinetic parameters, and/or biologic (pharmacodynamic) results.

VI. To describe the responses of this treatment combination.

OUTLINE: This is a multicenter, phase I, dose-escalation study. COHORT I: Patients receive oral dasatinib and oral lapatinib ditosylate once daily on days 1-28.

COHORT II: Patients receive oral dasatinib once daily on days 1 and 9-28 and oral lapatinib ditosylate once daily on days 2-28 of course 1. In all subsequent courses patients receive oral dasatinib and oral lapatinib ditosylate once daily on days 1-28.

In both cohorts courses repeat every 28 days, in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now unresectable and refractory to or refused all standard treatment for the disease
* Please contact study investigator and/or consult protocol document for specific details on laboratory criteria
* Ability to provide informed consent
* Willingness to return to Mayo Clinic for follow up
* Life expectancy >= 12 weeks
* Negative serum pregnancy test done =< 7 days prior to registration for women of childbearing potential only
* Echocardiogram with ejection fraction > 50%
* ECOG performance status (PS) 0-2
* Able to swallow pills whole (patients with feeding tubes may be eligible if whole pills can be taken and tolerated through the feeding tube)
* Willingness to provide the biologic specimens as required by the protocol for Cohort II, (MTD) patients only

Exclusion Criteria:

* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Pregnant women
* Any of the following prior therapies: chemotherapy =< 4 weeks prior to registration; mitomycin C/nitrosoureas =< 6 weeks prior to registration; immunotherapy =< 4 weeks prior to registration; biologic therapy =< 4 weeks prior to registration
* Patients who have been treated with Avastin, Herceptin, or Erbitux are eligible if last treatment is >= 4 weeks; molecularly targeted agents (erlotinib, sunitinib, sorafenib, gefitinib, imatinib) =< 4 weeks prior to registration; radiation therapy =< 4 weeks prior to registration; radiation to > 25% of bone marrow
* CNS metastases that are not stable for at least 4 weeks prior to registration based on imaging, clinical assessment, and use of steroids
* Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study and until 4 weeks following study
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation)
* Current therapy with a CYP3A4 inhibitor or inducer
* Known standard therapy for the patient's disease that is not refractory to treatment that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled pleural or pericardial effusion of any grade
* Uncontrolled angina, congestive heart failure or MI within 6 months prior to registration
* Diagnosed congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Subjects with potassium or magnesium that are not within normal limits and cannot be corrected prior to registration
* New York Heart Association classification III or IV
* Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Ongoing or recent (=< 3 months prior to registration) significant gastrointestinal bleeding
* Prophylactic use of colony-stimulating factors during the study is not allowed
* Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* G.I conditions that may interfere with drug absorption such as Ulcerative Colitis, Crohn's Disease, and Short Bowel Syndrome
* Active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator's assessment)
* Nursing women
* Uncontrolled infection
* Seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2014-12-18 (Actual); Study Completion 2014-12-18 (Actual)

PRIMARY OUTCOMES:
Adverse events profile
Toxicity profile per NCI CTCAE v3.0
Response profile | Every 4 weeks
Time until any treatment-related toxicity, time until treatment-related grade 3+ toxicity, and time until hematologic nadirs (WBC, ANC, platelets)
Time to progression and time to treatment failure
Laboratory correlates

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota